CLINICAL TRIAL: NCT05791578
Title: Corresponding Author
Brief Title: Relationship Obsessive Beliefs and Thought Control
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Meltem puşuroğlu, assistant professor doctor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: RTEuniversity
Record Dates: First submitted 2023-01-30; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Obsessive Thoughts
Keywords: panic disorder; generalized anxiety disorder
MeSH Terms: conditions — Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obsessive beliefs and thought control have been mostly investigated in obsessive-compulsive disorder in the literature. However, there is an increasing body of literature indicating that obsessive beliefs and thought control also play a role in the development of other anxiety disorders. In the study, investigators hypothesised that obsessive beliefs and thought control are effective in generalised anxiety disorder and panic disorder and increase anxiety symptoms and aimed to investigate the accuracy of this hypothesis.

DETAILED DESCRIPTION:
Obsessive beliefs are considered as a compulsive thought system in the cognitive model of obsessive-compulsive disorder. Obsessive beliefs are analysed under six main headings. These are control of thoughts, intolerance of uncertainty, exaggerated perception of responsibility, overemphasis of thoughts, exaggerated perception of threat and perfectionism. Although it is thought to play a role in the development of obsessions, it can sometimes be seen independent of obsessions . This dysfunctional distorted thought system sometimes turns into unnecessary threat perception and may pave the way for mental illnesses in the individual. When these distorted cognitive thoughts come to the mind, the person has an excessive mental effort to control the thoughts. As much as the thoughts cause distress, the endeavour to control the thoughts may cause mental distress in the person. Although all of these dysfunctional thoughts are associated with an obsession, the effect of thought control and obsessive beliefs on other mental illnesses has recently been investigated. In particular, perfectionism and increased threat perception have been associated with anxiety disorders as well as obsessions . Obsessive beliefs have often been associated with obsessive-compulsive disorder. However, there are similarities in the cognitive schemas of obsessive-compulsive disorder and anxiety disorders. Anxiety disorders are characterised by a vague state of anxiety and accompanying physical symptoms. Patients with anxiety disorders may be hypersensitive to some feelings and thoughts. Anxiety attacks may be triggered by exaggerated threat perception in obsessive beliefs. In addition, intolerance of uncertainty is also associated with anxiety disorders. Cognitive distortions have a role in the development of both obsessive-compulsive disorder and anxiety disorders . Obsessive beliefs and thought control have been mostly associated with obsessive-compulsive disorder in the literature. However, it has recently been thought that these dysfunctional compulsive thoughts and the distress experienced to control these thoughts are the cognitive basis of all anxiety disorders. Information on this subject is limited in the literature. Our study aims to contribute to the literature on this subject.

ELIGIBILITY:
Inclusion Criteria:

* with panic disorder patient and generalized anxiety disorder
* no other psychiatric illness such as alzheimer, mental retardation, parkinson disease
* had academic capacity for filling the scales
* no taking any drugs
* being age 18-65
* giving consent to be involved in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: with panic disorder patient and generalized anxiety disorder patient
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
The study will include healthy controls, patients with panic disorder and patients with anxiety disorder. 3 groups will be formed and obsessive beliefs scale and thought control scale will be applied to the groups. | 3 months
  Obsessive beliefs and will be applied in patients with panic disorder and anxiety disorder. scale results will be evaluated statistically. the hypothesis of the study is that obsessive beliefs scale scores will be higher in the patient group. The mentioned scales are the scales used for diagnosis in psychiatry. the answers have a score and a numerical value is obtained by adding the scores. the lowest score that can be obtained from the obsessive beliefs scale is 44 and the highest score is 208. higher scores on the scale are negative and mean more obsessive beliefs
The study will include healthy controls, patients with panic disorder and patients with anxiety disorder. 3 groups will be formed and obsessive beliefs scale and thought control scale will be applied to the groups. | 3 months
  thought control scale will be applied in patients with panic disorder and anxiety disorder. scale results will be evaluated statistically. the hypothesis of the study is that thought control scale scores will be higher in the patient group. The mentioned scales are the scales used for diagnosis in psychiatry. the answers have a score and a numerical value is obtained by adding the scores.. the lowest score that can be obtained from the thought control scale is 30 and the highest is 120. increasing scores were evaluated negatively. it is associated with more difficult thought control.

CONTACTS AND LOCATIONS:
Locations (1):
- RTE University, Rize, Turkey (Türkiye)